CLINICAL TRIAL: NCT05459610
Title: Development and Validation of an Artificial Intelligence System for Automatic Evaluation of the Extent of Intestinal Metaplasia
Brief Title: Automatic Evaluation of the Extent of Intestinal Metaplasia With Artificial Intelligence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Other Study IDs: 2022SDU-QILU-109
Record Dates: First submitted 2022-07-08; First posted 2022-07-15 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Intestinal Metaplasia of Gastric Mucosa; Artificial Intelligence; Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group for training the algorithm: This group of images is used for training the algorithm of the artificial intelligence
- group for testing the algorithm: This group of images is used for testing the algorithm of the artificial intelligence

SUMMARY:
Gastric intestinal metaplasia(GIM) is an important stage in the gastric cancer(GC). With technical advance of image-enhanced endoscopy (IEE), studies have demonstrated IEE has high accuracy for diagnosis of GIM. The endoscopic grading system (EGGIM), a new endoscopic risk scoring system for GC, have been shown to accurately identify a wide range of patients with GIM. However, the high diagnostic accuracy of GIM using IEE and EGGIM assessments performed all require much experience, which limits the application of EGGIM. The investigators aim to design a computer-aided diagnosis program using deep neural network to automatically evaluate the extent of IM and calculate the EGGIM scores.

DETAILED DESCRIPTION:
Globally, gastric cancer is the fifth most prevalent malignancy and the third leading cause of cancer mortality. Gastric intestinal metaplasia (GIM) is an intermediate precancerous gastric lesion in the gastric cancer cascade. Studies have shown that the 5-year cumulative incidence of gastric cancer in IM patients ranges from 5.3% to 9.8% . With technical advance of image-enhanced endoscopy (IEE), studies have demonstrated IEE has high accuracy for diagnosis of GIM. The endoscopic grading system (EGGIM), a new endoscopic risk scoring system for GC, have been shown to accurately identify a wide range of patients with GIM. However, The high diagnostic accuracy of GIM using IEE and EGGIM assessments performed all require much experience, which limits the application of EGGIM. The investigators aim to design a computer-aided diagnosis program using deep neural network to automatically evaluate the extent of IM and calculate the EGGIM scores.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-80 years who undergo the IEE examination

Exclusion Criteria:

* patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in gastroscopy
* patients with previous surgical procedures on the stomach
* patients who refuse to sign the informed consent form

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients who receive the IEE examination and screened that fulfill the eligibility criteria at Qilu Hospital, Shandong University will be enrolled into the study
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
The specificity of AI model to assess the degree of intestinal metaplasia in an endoscopic picture | 2 years
  The specificity of AI model to assess the degree of intestinal metaplasia in an endoscopic picture
The accuracy of AI model to assess the degree of intestinal metaplasia in an endoscopic picture | 2 years
  The accuracy of AI model to assess the degree of intestinal metaplasia in an endoscopic picture
The sensitivity of AI model to assess the degree of intestinal metaplasia in an endoscopic picture | 2 years
  The sensitivity of AI model to assess the degree of intestinal metaplasia in an

SECONDARY OUTCOMES:
Accuracy of the experienced endoscopists to assess the degree of intestinal metaplasia | 2 years
  Accuracy of the experienced endoscopists to assess the degree of intestinal metaplasia in an endoscopic picture
Accuracy of the inexperienced endoscopists to assess the degree of intestinal metaplasia | 2 years
  Accuracy of the inexperienced endoscopists to assess the degree of intestinal metaplasia in an endoscopic picture
Inter-observer agreement among experienced endoscopists in identifying the degree of intestinal metaplasia | 2 years
  Inter-observer agreement among experienced endoscopists in identifying the degree of intestinal metaplasia in an endoscopic picture
Inter-observer agreement among inexperienced endoscopists in identifying degree of intestinal metaplasia | 2 years
  Inter-observer agreement among inexperienced endoscopists in identifying degree of intestinal metaplasia in an endoscopic picture

CONTACTS AND LOCATIONS:
Overall Officials: yanqing Li, MD, PHD, Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastrology, QiLu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No